CLINICAL TRIAL: NCT01423058
Title: A Phase I/II, Open-Label Study Evaluating Twice-Daily Administration of CYT387 in Primary Myelofibrosis or Post-Polycythemia Vera or Post-Essential Thrombocythemia Myelofibrosis
Brief Title: Safety Study Evaluating Twice-Daily Administration of Momelotinib in Primary Myelofibrosis or Post-Polycythemia Vera or Post-Essential Thrombocythemia Myelofibrosis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sierra Oncology LLC - a GSK company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YM387-II-02
Record Dates: First submitted 2011-07-07; First posted 2011-08-25 (Estimated); Last update posted 2019-02-04 (Actual); Status verified 2019-01

CONDITIONS: Primary Myelofibrosis; Post-Polycythemia Vera; Post-Essential Thrombocythemia Myelofibrosis
MeSH Terms: conditions — Primary Myelofibrosis | interventions — N-(cyanomethyl)-4-(2-((4-(4-morpholinyl)phenyl)amino)-4-pyrimidinyl)benzamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Momelotinib (Experimental)
  Interventions: Drug: Momelotinib

INTERVENTIONS:
Drug: Momelotinib — In the Part I dose-escalation phase of the study, subjects will be assigned to dose levels in successive cohorts starting with a dose in the first cohort of 200 mg BID (twice daily with doses taken approximately 12 hours apart. Doses will be escalated by 50 mg BID in successive cohorts of 3 subjects per dose level. Subjects will be evaluated weekly for the first cycle, every 2 weeks during cycle 2, then monthly for 4 cycles for a total of 6 cycles.
  In the dose confirmation phase of the study (Part 2), subjects will be evaluated every 2 weeks during the first treatment cycle, and then monthly for 5 cycles for a total of 6 cycles.
  Other Names: CYT387

SUMMARY:
The myeloproliferative neoplasms (MPN), most notably polycythemia vera (PV), essential thrombocythemia (ET), and primary myelofibrosis (PMF) are a diverse but inter-related suite of clonal disorders of pluripotent hematopoietic stem cells (Tefferi et al., 2008). The MPN share a range of biological, pathological, and clinical features including the relative overproduction of one or more cells of myeloid origin, growth factor independent colony formation in vitro, marrow hypercellularity, extramedullary hematopoiesis, spleno- and hepatomegaly, and thrombotic and/or hemorrhagic diatheses (Tefferi et al., 2005).

This is a multi-centre, open-label, non-randomized, dose-escalation study, to be conducted in two phases: a dose-escalation phase (Part 1), to determine the safety and tolerability of momelotinib (CYT387), and to identify a therapeutic dose for the expanded cohort; and a dose-confirmation phase (Part 2), which will be a cohort expansion at or below the MTD of momelotinib.

In the Part I dose-escalation phase of the study, subjects will be assigned to dose levels in successive cohorts starting with a dose in the first cohort of 200 mg BID (twice daily with doses taken approximately 12 hours apart). Doses will be escalated by 50 mg BID per cohort until dose-limiting toxicities are observed. The dose level at which ≥2 of 6 subjects develop a first cycle dose-limiting toxicity (DLT) is defined as the DLT level. The maximum tolerated dose (MTD) is defined as the dose level below the DLT level. New dose levels may begin accrual only if all subjects at the current dose level have been observed for a minimum of 28 days from the first day of treatment. The dose level chosen for study in the dose confirmation phase of the study will be the MTD or a lower dose shown to have significant clinical activity (efficacy) as determined by the safety review committee. Subjects will be evaluated weekly for the first cycle, every 2 weeks during cycle 2, then monthly for 4 cycles for a total of 6 cycles.

In the dose-confirmation phase of the study, approximately fifty (50) subjects will be treated at the MTD or at a lower dose shown to have significant clinical activity (efficacy) as chosen by the Safety Review Committee. In the dose confirmation phase of the study subjects will be evaluated every 2 weeks during the first treatment cycle, and then monthly for 5 cycles for a total of 6 cycles.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of PMF or post-ET/PV MF as per revised World Health Organization (WHO) criteria (Section 16.4, Appendix 3).
* High-risk or Intermediate-2 risk MF (as defined by the International Prognostic Scoring System [IPSS]; Section 16.6, Appendix 5); or Intermediate-1 risk MF (IPSS) associated with symptomatic splenomegaly/hepatomegaly and/or unresponsive to available therapy.
* Must be at least 18 years of age with life expectancy of ≥ 12 weeks.
* Must be able to provide informed consent and be willing to sign an informed consent form.
* Must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1 or 2 (Section 16.3, Appendix 2).
* Must have evidence of acceptable organ function within 7 days of initiating study drug as evidenced by the following:
* AST or ALT less than or equal 2.5 x upper limit of normal (ULN) (or less than or equal to 5 x ULN if in the investigator's opinion the elevation is due to extramedullary hematopoiesis)
* Direct Bilirubin less than or equal to 2.0 x ULN
* Serum creatinine less than or equal to 2.5 x ULN
* Absolute neutrophil count ≥ 500/µL
* Platelet count ≥ 50,000/µL
* Females of childbearing potential must have a negative pregnancy test within 4 days of initiating study drug.

Exclusion Criteria:

* Any chemotherapy (e.g., hydroxyurea), immunomodulatory drug therapy (e.g., thalidomide), immunosuppressive therapy, corticosteroids >10 mg/day prednisone or equivalent, or growth factor treatment (e.g., erythropoietin) within 14 days prior to initiation of study drug.
* Incomplete recovery from major surgery within four weeks of study entry.
* Radiation therapy within four weeks of study entry.
* Women of childbearing potential, unless surgically sterile for at least 3 months (i.e., hysterectomy), OR postmenopausal for at least 12 months (FSH > 30 U/mL), OR unless they agree to take appropriate precautions to avoid pregnancy (with at least 99% certainty) from screening through end of study. Permitted methods for preventing pregnancy must be communicated to study subjects and their understanding confirmed.
* Men who partner with a woman of childbearing potential, unless they agree to take appropriate precautions to avoid pregnancy (with at least 99% certainty) from screening through to the end of study. Permitted methods for preventing pregnancy must be communicated to study subjects and their understanding confirmed.
* Females who are pregnant or are currently breastfeeding.
* Known positive status for HIV.
* Positive serologic testing for hepatitis B (HBsAg and HBcAb total) and hepatitis C (anti-HCV)
* Diagnosis of another malignancy unless free of disease for at least three years following therapy with curative intent. Patients with early-stage basal cell or squamous cell skin cancer, cervical intraepithelial neoplasia, cervical carcinoma in situ or superficial bladder cancer may be eligible participate at the Investigator's discretion.
* Any acute active infection.
* Cardiac dysrhythmias requiring treatment, or prolongation of the QTc (Fridericia) interval to >480 at pre-study screening, unless attributable to pre-existing bundle branch block.
* Presence of ≥ grade 2 peripheral neuropathy.
* Uncontrolled congestive heart failure (New York Heart Association Classification 3 or 4), uncontrolled or unstable angina, myocardial infarction, cerebrovascular accident, or pulmonary embolism within 3 months prior to initiation of study drug.
* Uncontrolled intercurrent illness or any concurrent condition that, in the Investigator's opinion, would jeopardize the safety of the patient or compliance with the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2011-08; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
To determine the safety of momelotinib by characterization and relationship of adverse events, affects on vital signs and laboratory parameters, and QTc intervals as measured by electrocardiogram (ECG) | 6 months
To determine maximum tolerated dose of momelotinib by characterization of Dose Limiting Toxicities | 6 months
To confirm the half-life of momelotinib by pharmacokinetic analyses | 6 months
To determine the efficacy of momelotinib by evaluation of spleen and liver size, disease related constitutional symptoms, transfusion dependence and anemia response. | 6 months

SECONDARY OUTCOMES:
To determine the effect of momelotinib on JAK2V617F mutant allele burden via Polymerase Chain Reaction (PCR) analyses | 6 months
To determine the effect of momelotinib on plasma levels of inflammatory, fibrogenic and angiogenic cytokines via Enzyme-Linked Immunosorbent Assay (ELISA) | 6 months
To determine the effect of momelotinib on bone marrow or peripheral blood cytogenetic findings | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Mark Kowalski, M.D., Study Director — YM Biosciences Inc.
Locations (6):
- United States (4):
  - Mayo Clinic, Scottsdale, Arizona
  - Mayo Clinic, Jacksonville, Florida
  - MD Anderson Cancer Center, The University of Texas, Houston, Texas
  - Huntsman Cancer Institute at the University of Utah, Salt Lake City, Utah
- Canada (2):
  - Princess Margaret Hospital, Toronto, Ontario
  - Jewish General Hospital, Montreal, Quebec

REFERENCES:
- [Derived] Gupta V, Mesa RA, Deininger MW, Rivera CE, Sirhan S, Brachmann CB, Collins H, Kawashima J, Xin Y, Verstovsek S. A phase 1/2, open-label study evaluating twice-daily administration of momelotinib in myelofibrosis. Haematologica. 2017 Jan;102(1):94-102. doi: 10.3324/haematol.2016.148924. Epub 2016 Sep 15. PMID 27634203